CLINICAL TRIAL: NCT05852678
Title: The Cantabria Cohort, a Protocol for a Population-based Cohort in Northern Spain
Brief Title: A Population-based Cohort in Northern Spain
Acronym: COHORTE
Status: Recruiting | Type: Observational
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Other Study IDs: COHORTE CANTABRIA; 2021.057 (Registry Identifier: cohorte)
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-04

CONDITIONS: Chronic Disease
Keywords: Lifestyle; Socio-economic factors; Biobank; Big data; Precision medicine; Longitudinal study
MeSH Terms: conditions — Chronic Disease | interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be used to measure conventional analytical parameters as well as serological markers of viral infection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient registry: The Cantabria Cohort will recruit 40,000-50,000 residents aged 40-69 years at baseline
  Interventions: Other: cohort

INTERVENTIONS:
Other: cohort — The Cantabria Cohort will recruit 40,000-50,000 residents aged 40-69 years at baseline

SUMMARY:
Cantabria Cohort stems from a research and action initiative lead by researchers from Valdecilla Research Institute (IDIVAL), Marqués de Valdecilla University Hospital and University of Cantabria, supported by the regional Goverment. Its aim is to identify and follow up a cohort that would provide information to improve the understanding of the etiology and prognosis of different acute and chronic diseases. The Cantabria Cohort will recruit between 40,000-50,000 residents aged 40-69 years at baseline, representing 10-20% of the target population. Currently, more than 22,000 volunteers have been enrolled. All participants will be invited for a re-assessment every three years, while the overall duration is planned for twenty years. The repeated collection of biomaterials combined with broad information from participant questionnaires, medical examinations, actual health system records and other secondary public data sources is a major strength of its design, which will make it possible to address biological pathways of disease development, identify new factors involved in health and disease, design new strategies for disease prevention, and advance precision medicine. It is conceived to allow access to a large number of researchers worldwide to boost collaboration and medical research.

DETAILED DESCRIPTION:
Recent reports have shown that non-communicable diseases, especially cardiovascular and metabolic diseases, were the main cause of morbi-mortality in Spain in 2019. Therefore, risks factors related to lifestyle, behavior and environment are placing a heavy burden on the Spanish population's health. At the same time, incidence of these diseases and an aging population threaten the sustainability of the Spanish universal health system. That stated, preventive, predictive and personalized medicine are urgently needed; to achieve such an aim, extensive data and knowledge will be fundamental.

Long-term follow-up cohort studies have played a crucial role in understanding modifiable factors associated with the development of chronic disease. In the early 1950s, initial results from the Framingham Health Study were published, beginning a new era in epidemiology . Large prospective cohort studies have established themselves as the most appropriate epidemiological design for research in the field of multimorbidity in real-life conditions. Over the last decades, the number of large prospective cohorts have increased.

The Framingham Health study selected its study population from a well-defined geographic area, the city of Framingham (Massachusetts, USA). This same strategy was carried out in Europe. One of the most remarkable examples was that of the European Prospective Investigation into Cancer and Nutrition (EPIC), which was an initiative of the International Agency for Research on Cancer (IARC). More recently, national cohort studies have been developed.

In Spain, several efforts have been undertaken to establish prospective, population-based cohorts. However, to date, long-term, population-based and multipurpose studies covering a specific territory have not been attemped. Conversely, a national cohort study has just been launched. Health system management in Spain takes place at the regional (autonomous community) level, which in practice results in 17 autonomous health systems within Spain.

In this context, the Cantabria Cohort was launched in late 2020 and it includes residents in Cantabria, an autonomous community located in northern Spain. Cantabria covers an area of 5,330 km², hosting a total population of 584,507 inhabitants, 45% living in the region's capital. Moreover, the Cantabrian Public Health System is organized into 42 health areas for primary care. It has four hospitals; the Hospital Universitario Marqués de Valdecilla (HUMV) is the tertiary and referenced hospital in the region. This center helps implement large-scale studies, reducing the necessity of coordination among different institutions and procedures. Further, due to the widespread COVID-19 vaccination campaign in 2021, a huge effort to integrate multiple public databases and update contact information of the population has facilitated the start of the project. Cantabria Cohort stems from a research and action initiative to improve the regional health system and advance the health-related Sustainable Development Goals. The present paper describes the design and implementation of the Cantabria Cohort and the processes related to the biological sample collection and data acquisition. It also provides an overview of the governing board, quality assurance, and legal and ethical aspects, as well as future research opportunities and cooperation.

ELIGIBILITY:
Inclusion Criteria:

* Participants between 40-69 years of age
* Participants who sign the informed consent form
* Participants legally residing in Cantabria

Exclusion Criteria:

* Participants under 40 years of age and over 69 years of age
* Participants not signing the informed consent form
* Participants not legally residing in Cantabria

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents in the autonomous community of Cantabria
Sampling Method: Non-Probability Sample
Enrollment: 22000 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2045-04-01 (Estimated); Study Completion 2045-04-01 (Estimated)

PRIMARY OUTCOMES:
Integration and use of real-world data to improve health research | 20 years
Identifying lifestyle risk factors and their involvement in chronic diseases | 20 years
Evaluation of geographic and socio-economic disparities in health and healthcare | 20 years
Assessing biomarkers for the early detection of diseases and disease risks | 20 years
Surveillance of viral hepatitis and HIV in Cantabria | 20 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Marques de Valdecilla, Santander, Spain